CLINICAL TRIAL: NCT01061177
Title: A Phase IIIb, Multicentre, Open-label Study of Nilotinib in Adult Patients With Newly Diagnosed Philadelphia Chromosome and/or BCR-ABL Positive CML in Chronic Phase
Brief Title: Nilotinib in Newly Diagnosed Adult Philadelphia Chromosome & /or BCR-ABL Positive Chronic Myeloid Leukaemia in Chronic Phase
Acronym: 'MACS1252
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107EIC01; 2009-017775-19 (EudraCT Number)
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2016-12

CONDITIONS: CML in Chronic Phase
Keywords: Leukemia; myeloid; myelogenous; chronic BCR-ABL positive; Nilotinib; Philadelphia chromosome; CML in chronic phase
MeSH Terms: conditions — Leukemia; Philadelphia Chromosome | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib (Experimental): This was a single-arm study; therefore all participants received nilotinib (AMN107) 300 mg bid given as two 150 mg capsules twice daily.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib was supplied by Novartis as 150 mg hard gelatin capsules in bottles. Nilotinib was dosed on a flat scale and not dosed by body weight. This form of supply was continued for all participants entered into the core study.
  Other Names: AMN107

SUMMARY:
This study will assess the efficacy and safety of nilotinib in adult patients with newly diagnosed Philadelphia chromosome positive/BCR-ABL positive chronic myeloid leukaemia in chronic phase. The aim of the study is to confirm the rates of complete molecular remission (CMR) of nilotinib in newly diagnosed CML chronic phase patients in a pan-European population using the EUTOS standardized laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of CP-CML with cytogenetic confirmation of Philadelphia (Ph) chromosome
* Ph negative cases or patients with variant translocations who are BCR-ABL positive in multiplex PCR are also eligible
* WHO performance status 0-2
* Laboratory assessments within normal limits
* Written informed consent prior to any study procedures being performed

Exclusion Criteria:

* Known impaired cardiac function
* History of acute or chronic pancreatitis
* Impaired gastrointestinal function or disease that may alter the absorption of study drug
* Concomitant medications with potential QT prolongation, or known to interact with CYP450 isoenzymes (CYP3A4, CYP2C9, and CYP2C8)
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding, or females of reproductive potential not employing an effective method of birth control. Female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Actual)
Dates: Start 2010-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (290):
- Austria (7):
  - Novartis Investigative Site, Wels, Austria
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (13):
  - Novartis Investigative Site, Aalst, Belgium
  - Novartis Investigative Site, Luxembourg, Luxembourg
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Verviers
  - Novartis Investigative Site, Yvoir
- Bulgaria (4):
  - Novartis Investigative Site, Pleven, Bulgaria
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Croatia (2):
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zagreb
- Czechia (4):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Hradec Králové, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
- Denmark (3):
  - Novartis Investigative Site, Aarhus C
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense C
- Novartis Investigative Site, Tartu, Estonia
- Finland (2):
  - Novartis Investigative Site, HUS Helsinki
  - Novartis Investigative Site, Oulu
- France (54):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Saint-Denis, France / La Reunion
  - Novartis Investigative Site, Angers, France
  - Novartis Investigative Site, Dunkirk, France
  - Novartis Investigative Site, Monte-Carlo, Principauté de Monaco
  - Novartis Investigative Site, Aix-en-Provence
  - Novartis Investigative Site, Amiens Cedex1
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Blois
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Chalon-sur-Saône
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Le Coudray
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lens
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Mâcon
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Montfermeil
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pau
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Pringy
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Roubaix
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Brieuc
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Saint-Quentin
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Troyes
- Germany (68):
  - Novartis Investigative Site, Eschweiler, Germany
  - Novartis Investigative Site, Kiel, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt (Oder)
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herrsching am Ammersee
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Landshut
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lemgo
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Mutlangen
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Paderborn
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Sindelfingen
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Traunstein
  - Novartis Investigative Site, Triberg
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Viersen
  - Novartis Investigative Site, Weilheim
  - Novartis Investigative Site, Wendlingen
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zella-Mehlis
- Greece (7):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Pátrai, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Italy (43):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Cuneo, CN
  - Novartis Investigative Site, Rossano, CS
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Livorno, LI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Nuoro, NU
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pesaro, PU
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Potenza, PZ
  - Novartis Investigative Site, Ravenna, RA
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Nocera Inferiore, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Taranto, TA
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Treviso, TV
  - Novartis Investigative Site, Ronciglione, VT
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Perugia
- Novartis Investigative Site, Riga, LV, Latvia
- Lithuania (3):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Netherlands (7):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Zwolle
- Norway (5):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Tromsø
  - Novartis Investigative Site, Trondheim
- Poland (6):
  - Novartis Investigative Site, Warsaw, Poland
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (3):
  - Novartis Investigative Site, Lisbon, Portugal
  - Novartis Investigative Site, Porto, Portugal
  - Novartis Investigative Site, Porto
- Romania (6):
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Bucharest, Romania
  - Novartis Investigative Site, Timișoara, Romania
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
- Slovakia (3):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Bratislava
- Slovenia (2):
  - Novartis Investigative Site, Celje
  - Novartis Investigative Site, Ljubljana
- Spain (23):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Ourense, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Murcia, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Zaragoza, Zaragoza
- Sweden (8):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Huddinge
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Switzerland (4):
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Geneva
- United Kingdom (6):
  - Novartis Investigative Site, Uxbridge, London
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Dudley
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford

REFERENCES:
- [Derived] Gullaksen SE, Skavland J, Gavasso S, Tosevski V, Warzocha K, Dumrese C, Ferrant A, Gedde-Dahl T, Hellmann A, Janssen J, Labar B, Lang A, Majeed W, Mihaylov G, Stentoft J, Stenke L, Thaler J, Thielen N, Verhoef G, Voglova J, Ossenkoppele G, Hochhaus A, Hjorth-Hansen H, Mustjoki S, Sopper S, Giles F, Porkka K, Wolf D, Gjertsen BT. Single cell immune profiling by mass cytometry of newly diagnosed chronic phase chronic myeloid leukemia treated with nilotinib. Haematologica. 2017 Aug;102(8):1361-1367. doi: 10.3324/haematol.2017.167080. Epub 2017 May 18. PMID 28522574
- [Derived] Thielen N, Richter J, Baldauf M, Barbany G, Fioretos T, Giles F, Gjertsen BT, Hochhaus A, Schuurhuis GJ, Sopper S, Stenke L, Thunberg S, Wolf D, Ossenkoppele G, Porkka K, Janssen J, Mustjoki S. Leukemic Stem Cell Quantification in Newly Diagnosed Patients With Chronic Myeloid Leukemia Predicts Response to Nilotinib Therapy. Clin Cancer Res. 2016 Aug 15;22(16):4030-8. doi: 10.1158/1078-0432.CCR-15-2791. Epub 2016 Mar 22. PMID 27006491

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ITT: intent to treat; b3a2 & b2a2 +ve are categories of BCR-ABL transcripts (BCR-ABL1 is an abnormal gene found in chronic myeloid leukemia and acute lymphoblastic leukemia patients; CyR (Ph+ Patients Only) = cytogenic response for Philadelphia positive patients only.
Period: Overall Study
Arm/Group | Nilotinib
Started | 1089
ITT_MR (b2a2 &/or b3a2 +ve Pts Only) | 1056
ITT_CyR (Ph+ Patients Only) | 983
Completed | 881
Not Completed | 208
Not completed — Adverse Event | 117
Not completed — Withdrawal by Subject | 27
Not completed — Disease progression | 17
Not completed — Protocol Violation | 11
Not completed — Lost to Follow-up | 9
Not completed — New cancer therapy | 9
Not completed — Abnormal laboratory values | 6
Not completed — Abnormal test procedure results | 4
Not completed — Administratie problems | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all participants who received at least one dose of study drug.
Arm/Group | Nilotinib
Number analyzed (Participants) | 1089
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (14.87)
Gender [Count of Participants; unit: Participants]
  Female | 447
  Male | 642
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucacian | 1045
  Black | 6
  Oriental | 5
  Native American | 2
  Other | 31
Weight at baseline [Mean (Standard Deviation); unit: Kg] | 77.47 (15.730)
ECOG performance score [Number; unit: Participants] — ECOG = Eastern Cooperative Oncology Group
  Participants
    No restrictions (0) | 867
    Only light work (1) | 199
    Only self care (2) | 21
    Limited self care (3) | 0
    Completely disabled (4) | 0
    Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Molecular Response (MR4^0) at 18 Months
Description: MR4^0 was defined as either (i) detectable disease ≤ 0.01% BCR-ABL ratio (international scale (IS)) with mean ABL transcripts ≥ 10 000 or (ii) undetectable disease in complementary deoxyribonucleic acid (cDNA) with ≥ 10 000 ABL transcripts.
Time Frame: at 18 months
Population: Intent-to-treat_Molecular (ITT_MR) analysis set was a subset of the ITT population including the patients with typical BCR-ABL transcript at screening.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1056
Percentage of Participants | 38.3

2. Secondary Outcome: Percentage of Participants Free From Progression to Accelerated Phase/Blast Crisis (AP/BC) at 12 and 24 Months
Description: The following events were considered disease progression to AP/BC: Death due to disease under study; AP, as defined by any of the following: ≥ 15% blasts in the peripheral blood or bone marrow, but < 30% blasts in both the peripheral blood and bone marrow, ≥ 30% blasts plus promyelocytes in peripheral blood or bone marrow, ≥ 20% basophils in the peripheral blood, Thrombocytopenia (< 100 × 109/L) that was unrelated to therapy, Evidence of clonal evolution, as determined by medical review with consensus of the SSMC/DMC.
  BC was defined as: ≥ 30% blasts in peripheral blood or bone marrow, Appearance of extramedullary involvement other than hepatosplenomegaly proven by biopsy.
Time Frame: at 12 and 24 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1089
Percentage of participants
  Pts free from progression to AP/BC at 12 months | 99.4
  Pts free from progression to AP/BC at 24 months | 99.4

3. Secondary Outcome: Rate of Event Free Survival at 12 and 24 Months
Description: EFS was defined as the time from the date of Day 1 (first treatment) + 1 day to the first occurrence of any of the following: Loss of complete hematologic response (CHR), Loss of CCyR, Death from any cause, Progression to the AP or BC of CML, Not achieving CHR up to 3 months (ie, 91 + 15 days), Not achieving CCyR up to 18 months (ie, 548 + 15 days), whichever is earlier.
Time Frame: at 12 and 24 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1089
Percentage of participants
  Percentage of participants with EFS at 12 months | 71.7
  Percentage of participants with EFS at 24 months | 69.1

4. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) at, as Well as by, 12 and 24 Months
Description: MMR was defined as BCR-ABL ratio (IS) ≤ 0.1% in a peripheral blood sample. BCR-ABL1 is an abnormal gene found in chronic myeloid leukemia (CML) and acute lymphoblastic leukemia (ALL). The chromosomal defect in the Philadelphia chromosome is a translocation, in which parts of two chromosomes, 9 and 22, swap places. The result is that a fusion gene is created by juxtapositioning the Abl1 gene on chromosome 9 to a part of the BCR ("breakpoint cluster region") gene on chromosome 22. Depending upon the breakpoints on the BCR gene, there are several forms of fusion proteins.
Time Frame: 12 months, 24 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1056
Percentage of participants
  at 12 months | 56.2
  at 24 months | 61.1
  by 12 months | 68.8
  by 24 months | 80.3

5. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) at, as Well as by, 12 and 24 Months
Description: CCyR parameters were defined as 0% Philadelphia positive (Ph+) metaphases. Loss of CCyR was defined as a patient exceeding the CCyR criteria (ie, > 0% Ph+ metaphases) at a subsequent visit after the patient had achieved CCyR.
Time Frame: 12 and 24 months
Population: The ITT_CyR population was a subset of the ITT population including the Ph+ patients at screening was considered. Patients who had either no metaphases recorded at screening bone marrow or only negative metaphases recorded at screening bone marrow but had Ph+ metaphases at any visits after screening were also part of this population.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 983
Percentage of participants
  at 12 months | 72.4
  at 24 months | 65.6
  By Month 12 | 82.5
  By Month 24 | 89.0

6. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR) at, as Well as by, 12 and 24 Months
Description: Major cytogenetic response (MCyR) parameters were defined as 0 to 35% Philadelphia positive (Ph+) metaphases.
Time Frame: 12 and 24 months
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 983
Percentage of participants
  at 12 months | 73.8
  at 24 months | 66.2
  by 12 months | 86.7
  by 24 months | 91.4

7. Secondary Outcome: Percentage of Participants Free From Progression to AP/BC With MR4^0 at 12 Months
Description: as for outcome 2
Time Frame: at 12 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 400
Percentage of participants | 100.0

8. Secondary Outcome: Percentage of Participants With Event Free Survival in Participants Achieving MR4^0 at 12 Months
Description: EFS was defined as the time from the date of Day 1 (first treatment) + 1 day to the first occurrence of any of the following: Loss of complete hematologic response (CHR), Loss of CCyR, Death from any cause, Progression to the AP or BC of CML, Not achieving CHR up to 3 months (i.e. 91 + 15 days).
Time Frame: at 12 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 400
Percentage of participants | 87.0

9. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 12 and 24 Months
Description: PFS was defined by the study protocol as the time from the date of start of study drug to the date of earliest progression to AP/BC, or the date of death from any cause.
Time Frame: 12 months, 24 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1089
Percentage of participants
  at 12 months | 99.2
  at 24 months | 99.0

10. Secondary Outcome: Rate of Molecular Response (MR4^0) at, as Well as by, 12 and 24 Months
Description: as for outcome 1
Time Frame: 12 and 24 months
Population: The ITT_MR population was a subset of the ITT population including the patients with typical BCR-ABL transcript at screening ie, b3a2 and/or b2a2 were considered. This population was referred to as ITT_MR.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1056
Percentage of participants
  at 12 months | 30.7
  at 24 months | 40.2
  by month 12 | 36.9
  by month 24 | 55.0

11. Secondary Outcome: Rate of Molecular Response (MR4^5) at, as Well as by, 12 and 24 Months
Description: MR4^5 was defined as either (i) detectable disease ≤ 0.0032% BCR-ABL ratio (IS) with mean ABL transcripts ≥ 32 000 or (ii) undetectable disease in cDNA with ≥ 32 000 ABL transcripts).
Time Frame: 12 and 24 months
Population: The ITT_MR population was a subset of the ITT population including the patients with typical BCR-ABL transcript at screening ie, b3a2 and/or b2a2 were considered.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1056
Percentage of participants
  at 12 months | 15.2
  at 24 months | 21.9
  by 12 months | 20.6
  by 24 months | 38.4

12. Secondary Outcome: Rate of Complete Hematologic Response (CHR) at, as Well as by, 12 and 24 Months
Description: CHR was defined as all of the following present for ≥ 4 weeks in the peripheral blood: WBC count < 10 x 109/L, Platelet count < 450 x 109/L, No circulating peripheral blood blasts, promyelocytes, myelocytes, or metamyelocytes in the peripheral blood, The presence of < 5% basophils, No evidence of disease-related symptoms and extramedullary disease, including spleen and liver. Loss of CHR was defined as the appearance of any of the following after having achieved a CHR confirmed by a second determination ≥ 4 weeks later (unless associated with progression to AP/BC or death, which was considered to be a confirmed loss of CHR event on its own): WBC count that increased to > 20.0 x 109/L, Platelet count that increased to ≥ 600 x 109/L, Any palpable spleen, defined as size of spleen below costal margin > 5 cm, Appearance of > 5% myelocytes plus metamyelocytes, or any promyelocytes or blasts in the peripheral blood.
Time Frame: 12 months, 24 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of prticipants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1089
Percentage of prticipants
  by Month 24 | 89.1
  at 12 months | 82.7
  at 24 months | 75.5
  by Month12 | 86.2

13. Secondary Outcome: Percentage of Participants With Overall Survival at 12 and 24 Months
Description: OS was defined as the time between the date of Day 1 (first treatment) and the date of death from any cause. Deaths which occurred after the 24-month time window and which were occasionally reported by some Investigators were excluded from the analysis. This is in agreement with the protocol stating that patients were to be followed for survival and progression to AP/BC up to 24 months after the participants treatment start.
Time Frame: 12 months, 24 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1089
Percentage of participants
  at 12 months | 99.6
  at 24 months | 98.9

14. Secondary Outcome: Rate of Molecular Response (MR4^0) by 18 Months
Description: MR4^0 was defined as either (i) detectable disease ≤ 0.01% BCR-ABL ratio (international scale (IS)) with mean ABL transcripts ≥ 10 000 or (ii) undetectable disease in complementary deoxyribonucleic acid (cDNA) with ≥ 10 000 ABL transcripts.
  BCR = Breakpoint Cluster Region gene/BCR gene product
  BCR-ABL is fusion gene formed from the ABL gene from chromosome 9 fusing with the BCR gene on chromosome 22, the gene product is BCR-ABL tyrosine kinase
Time Frame: by 18 months
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1056
Percentage of participants | 48.5

15. Secondary Outcome: Rate of Molecular Response (MR4^5) by 18 Months
Description: MR4^5 was defined as either (i) detectable disease ≤ 0.0032% BCR-ABL ratio (IS) with mean ABL transcripts ≥ 32 000 or (ii) undetectable disease in cDNA with ≥ 32 000 ABL transcripts).
  BCR = Breakpoint Cluster Region gene/BCR gene product
  BCR-ABL is fusion gene formed from the ABL gene from chromosome 9 fusing with the BCR gene on chromosome 22, the gene product is BCR-ABL tyrosine kinase
Time Frame: by 18 months
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 1056
Percentage of participants | 31.6

16. Secondary Outcome: Percentage of Participants With Progression Free Survival in Participants Achieving MR4^0 at 12 Months
Description: as for outcome 9
Time Frame: 12 months
Population: The intent-to-treat (ITT) population consisted of all patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 400
Percentage of participants
  at 12 months | 99.2
  at 24 months | 99.0

ADVERSE EVENTS:
Arm/Group | Nilotinib
Serious Adverse Events (participants affected / at risk) | 207/1089
Other Adverse Events (participants affected / at risk) | 841/1089
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=1089)
Anaemia (Blood and lymphatic system disorders) | 5
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Splenic infarction (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Acute coronary syndrome (Cardiac disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 4
Angina pectoris (Cardiac disorders) | 6
Angina unstable (Cardiac disorders) | 2
Aortic valve stenosis (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 13
Atrial flutter (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 7
Coronary artery stenosis (Cardiac disorders) | 1
Coronary artery thrombosis (Cardiac disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Myocardial ischaemia (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Thyroiditis subacute (Endocrine disorders) | 1
Conjunctival disorder (Eye disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatic disorder (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 6
Pancreatitis acute (Gastrointestinal disorders) | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chest pain (General disorders) | 1
Device dislocation (General disorders) | 1
Drug resistance (General disorders) | 1
Fatigue (General disorders) | 2
Localised oedema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 6
Soft tissue inflammation (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Gallbladder enlargement (Hepatobiliary disorders) | 1
Hepatic fibrosis (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Corneal abscess (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Phlebitis infective (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Rectal abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Viral pericarditis (Infections and infestations) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2
Exposure via father (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Sternal injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Blood pressure increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 3
Lipase increased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Cranial nerve disorder (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Hyperaesthesia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Motor neurone disease (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Occipital neuralgia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
VIIth nerve paralysis (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Depression suicidal (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Genital pain (Reproductive system and breast disorders) | 1
Genital swelling (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Hysterectomy (Surgical and medical procedures) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1
Aneurysm ruptured (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 2
Arterial disorder (Vascular disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Leriche syndrome (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=1089)
Anaemia (Blood and lymphatic system disorders) | 65
Thrombocytopenia (Blood and lymphatic system disorders) | 111
Abdominal pain (Gastrointestinal disorders) | 79
Abdominal pain upper (Gastrointestinal disorders) | 88
Constipation (Gastrointestinal disorders) | 65
Diarrhoea (Gastrointestinal disorders) | 93
Nausea (Gastrointestinal disorders) | 122
Vomiting (Gastrointestinal disorders) | 62
Asthenia (General disorders) | 97
Fatigue (General disorders) | 150
Nasopharyngitis (Infections and infestations) | 113
Alanine aminotransferase increased (Investigations) | 86
Blood bilirubin increased (Investigations) | 80
Lipase increased (Investigations) | 76
Hypophosphataemia (Metabolism and nutrition disorders) | 77
Arthralgia (Musculoskeletal and connective tissue disorders) | 96
Back pain (Musculoskeletal and connective tissue disorders) | 78
Muscle spasms (Musculoskeletal and connective tissue disorders) | 93
Myalgia (Musculoskeletal and connective tissue disorders) | 99
Headache (Nervous system disorders) | 163
Insomnia (Psychiatric disorders) | 55
Cough (Respiratory, thoracic and mediastinal disorders) | 56
Alopecia (Skin and subcutaneous tissue disorders) | 115
Dry skin (Skin and subcutaneous tissue disorders) | 93
Pruritus (Skin and subcutaneous tissue disorders) | 180
Rash (Skin and subcutaneous tissue disorders) | 233
Hypertension (Vascular disorders) | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.